CLINICAL TRIAL: NCT06303258
Title: Comparison of Generalized Versus Core Stabilization Antenatal Exercises For Lumbopelvic Pain In Pregnancy
Brief Title: Generalized Versus Core Stabilization Antenatal Exercises For Lumbopelvic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU Sharmeen Kanwar
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Low Back Pain; Pelvic Pain
MeSH Terms: conditions — Low Back Pain; Pelvic Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single (Outcomes Assessor)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Core Stabalization Exercises Group (Experimental): This Group will receive core stability exercises 3 sessions per week for 4 weeks and basic antenatal education.
  Interventions: Other: Core Stabalization Exercises
- Generalized Exercise Group (Experimental): This Group will receive generalized supervised antenatal exercises that are covered in three phases and basic antenatal education. There will be 3 sessions per week for 10weeks conducted for generalized antenatal exercises including Aerobics, Endurance and Pelvic Floor Muscle Training.
  Interventions: Other: Generalized Antenatal Exercises
- Control Group (No Intervention): Basic Antenatal Education for Lumbopelvic Pain Prevention

INTERVENTIONS:
Other: Core Stabalization Exercises — Low Intensity Warm Up Exercises Core Stabilization Exercises Cool Down Stretching Exercises
  Arms: Core Stabalization Exercises Group
Other: Generalized Antenatal Exercises — Low Intensity WarmUp Exercise Aerobic Training Endurance Training Pelvic Floor Muscle Training Cool Down Stretching Exercises
  Arms: Generalized Exercise Group

SUMMARY:
Core stability training has gained popularity as a fitness trend and is now being used in rehabilitation programs as well the patient adherence to this intervention has been low due to its complex nature, particularly pregnant females .Limited literature is available to present the effect of core stabilization exercises in comparison to the other handful simplified techniques and exercises This study compares two interventions for this particular condition to identify a feasible and enjoyable therapeutic intervention for the pregnant women who suffer Lumbopelvic Pain.

DETAILED DESCRIPTION:
This is a randomized control trial to compare the effects of core stabilization versus generalized antenatal exercises for lumbopelvic pain in pregnant women. Females meeting the inclusion and exclusion criteria will be divided into three groups by convenient sampling technique. A sample size of 48 females with 16 females in each group. Group A will be treated by core stability exercises and group B will be treated by generalized antenatal exercises and group C will receive basic antenatal education. Group A and B will have three treatment sessions per week for 4 weeks. Females will be evaluated at baseline and 2nd and 4th week . Females will be screened by Patricks faber test, piriformis /FAIR test, p4/posterior pelvic pain provocation test and assessed by visual analogue scale (VAS) and pregnant women quality of life questionnaire (QOL- GRAV).

ELIGIBILITY:
Inclusion Criteria:

* 2nd Trimester of Pregnancy
* Multigravida
* Patients having Lumbopelvic pain
* Working women and housewives

Exclusion Criteria:

* Hx of Metabolic Disease
* Hx of Pelvic Fracture and Surgery
* Radiculopathy
* Participants with absolute contraindications for the exercise

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 48 (Actual)
Dates: Start 2024-03-04 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Changes from Baseline to 2nd week
  It is a numeric rating scale from 0 to 10 where 0 represents "no pain" and 10 represents the "worst possible pain.it is used to rate the pain intensity in patients
Visual Analogue Scale (VAS) | Changes from 2nd week to 4th week
  It is a numeric rating scale from 0 to 10 where 0 represents "no pain" and 10 represents the "worst possible pain.it is used to rate the pain intensity in patients
Pregnant women's quality of life questionnaire (QOL-GRAV) | Changes from Baseline to 2nd week
  Nine items make up the scale that allows individuals to describe their individual experiences with pregnancy's quality of life. It had a greater internal consistency than 0.7. A 5-point Likert scale (ranging from not at all [0] to totally [4]) was used to rate each item. The final three questions-7, 8 and 9-are scored in reverse.
Pregnant women's quality of life questionnaire (QOL-GRAV) | Changes from 2nd week to 4th week
  Nine items make up the scale that allows individuals to describe their individual experiences with pregnancy's quality of life. It had a greater internal consistency than 0.7. A 5-point Likert scale (ranging from not at all [0] to totally [4]) was used to rate each item. The final three questions-7, 8 and 9-are scored in reverse.

CONTACTS AND LOCATIONS:
Overall Officials: Huma Riaz, PHD, Principal Investigator — Riphah International University
Locations (1):
- Tehsil Headquarter Hospital Raiwind, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sklempe Kokic I, Ivanisevic M, Uremovic M, Kokic T, Pisot R, Simunic B. Effect of therapeutic exercises on pregnancy-related low back pain and pelvic girdle pain: Secondary analysis of a randomized controlled trial. J Rehabil Med. 2017 Mar 6;49(3):251-257. doi: 10.2340/16501977-2196. PMID 28233012
- [Background] Stuge B. Evidence of stabilizing exercises for low back- and pelvic girdle pain - a critical review. Braz J Phys Ther. 2019 Mar-Apr;23(2):181-186. doi: 10.1016/j.bjpt.2018.11.006. Epub 2018 Nov 17. PMID 30471967
- [Background] Varela-Esquivias A, Diaz-Martinez L, Avendano-Badillo D. [Efficacy of lumbopelvic stabilization exercises in patients with lumbalgia]. Acta Ortop Mex. 2020 Jan-Feb;34(1):10-15. Spanish. PMID 33230993
- [Background] Leonard JH, Paungmali A, Sitilertpisan P, Pirunsan U, Uthaikhup S. Changes in Transversus Abdominis Muscle Thickness after Lumbo-Pelvic Core Stabilization Training among Chronic Low Back Pain Individuals. Clin Ter. 2015;166(5):e312-6. doi: 10.7417/T.2015.1884. PMID 26550815